CLINICAL TRIAL: NCT02322060
Title: Ovarian Tissue Cryopreservation and Auto-transplantation for in Vitro Activation of Dormant Follicles for Patients with Primary Ovarian Insufficiency
Brief Title: In Vitro Activation of Dormant Follicles for Patients with Primary Ovarian Insufficiency
Acronym: IVADFPOI
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Stanford University (Other); St. Marianna University School of Medicine (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-IVA
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: In Vitro Activation; Dormant Follicle; Primary Ovarian Insufficiency; Ovarian Resistance Syndrome
Keywords: IVA, ovary tissue grafting, POI, ORS
MeSH Terms: conditions — Primary Ovarian Insufficiency; Acidemia, isovaleric; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum, ovary tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary ovarian insufficiency: Primary ovarian insufficiency (POI; also known as premature ovarian failure/dysfunction/insufficiency or premature menopause) is characterised by amenorrhoea, sex hormone (oestrogen, progesterone and testosterone) deficiency and elevated gonadotrophins levels in a woman aged more than two standard deviations below the mean age of menopause estimated for her reference population. POI is defined as a disorder in ovarian function in any woman before the age of 40 years, irrespective of the cause.
  In our study, we mainly recruit POI patients who also desire to have a baby of their own.
  Interventions: Procedure: Ovariotomy; Procedure: Activate dormant follicles; Procedure: Ovary tissue transplantation; Procedure: Ovarian superficial cut
- Ovarian resistance syndrome: We currently also include patients diagnosed with Ovarian resistance syndrome, which means that follicles exist, but do not response to FSH.
  Interventions: Procedure: Ovariotomy; Procedure: Activate dormant follicles; Procedure: Ovary tissue transplantation; Procedure: Ovarian superficial cut

INTERVENTIONS:
Procedure: Ovariotomy — Remove one ovary (maybe both ovaries depending on the condition) by laparoscopic surgery or by laparotomy in some cases.
Procedure: Activate dormant follicles — Cut ovary into small cubes, which are then cultured with medium containing BPV(pic), a PTEN inhibitor, and 740YP, an activator of phosphoinositol 3 kinase, to activate dormant follicles for 2 days before transplantation.
Procedure: Ovary tissue transplantation — After extensive washing to remove drugs, the ovary cubes are transplanted beneath the membrane of both Fallopian tubes and the remaining ovary under laparoscopic surgery.
Procedure: Ovarian superficial cut — Superficial cut of the ovarian cortex by laparoscopy or laparotomy

SUMMARY:
In this study, the investigators used the newly developed technique i.e. in vitro activation of dormant follicles (IVA) to promote ovarian follicle growth much more efficiently than natural, in vivo process for women with Primary Ovarian Insufficiency (POI).Firstly, the investigators remove one ovary under laparoscopic surgery. Then, we dissect ovarian cortex from the ovarian medulla. The ovarian cortex is cut into small cubes and cultured with medium containing drugs to activate dormant follicles. After 2 days of culture, the ovarian cubes are transplanted mainly beneath the membrane of Fallopian tubes under laparoscopic surgery. The ovarian cortex could be cryopreserve for future re-transplantation and in some cases, for convenience to arrange second surgery. Once frozen, the ovary can be preserved semipermanently. After transplantation, patients receive ultrasound monitoring together with measurement of serum hormone levels for 10-12 months. If growing follicles are detected, follicle growth is stimulated by injection of hormones (gonadotropins). Using the same "ovum pick up" approach used in IVF (in vitro fertilization), we pick up oocytes from the follicles and fertilize them. Fertilized eggs are cultured and then cryopreserved for future embryo transfer.

Currently, we recurit patients diagnosed with POI, or Ovarian resistance syndrome (ORS). The procedure can also be: Only superficial cut of the ovarian cortex by laparoscopy or laparotomy, without taking ovary outside or cultured with medium.

DETAILED DESCRIPTION:
I: Former IVA

1. Remove one ovary (maybe both ovaries depending on the condition) is performed by laparoscopic surgery. (Depending on the condition of patients, the investigators remove both ovaries to increase a chance to obtain residual follicles. Also, in some cases, the investigators need to perform laparotomy, i.e. open surgery, depending on the patient's condition).
2. Quickly dissect ovarian cortex from the ovarian medulla and cut into small stripes. Histological analyses are performed using small parts of the ovarian stripes to find residual follicles.
3. Optional: Cryopreserve the ovarian stripes by a vitrification method. Two days before the day of reimplantation, thaw the ovarian stripes.
4. The ovarian stripes are cut into small cubes (1 x1 mm2). The ovarian cubes are cultured with medium containing drugs to activate dormant follicles for 2 days before transplantation. After washing, the cubes are transplanted beneath the membrane of both Fallopian tubes and the remaining ovary under laparoscopic surgery.
5. Monitor follicle growth by ultrasound and serum hormone assays. Once follicles reach >16 mm in diameter, patients receive hCG, followed by egg retrieval in ~36 hours. Then the investigators will perform intracytoplasmic sperm injection (ICSI) using the husband's sperm. When embryos reached the four-cell stage, they were cryopreserved, waiting for frozen-thaw embryo transfer.

II Current procedure:

Only superficial cut of the ovarian cortex by laparoscopy or laparotomy, without taking ovary outside or cultured with medium.

ELIGIBILITY:
Inclusion Criteria:

* Married women (18-39) diagnosed with POI/ORS
* With both ovaries present
* With normal uterine cavity
* Healthy and can stand surgery

Exclusion Criteria:

* Any one that does not meet the inclusion criteria

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women diagnosed with POI/ORS who also want to get pregnant by IVF/ICSI-ET with their own oocyte.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2021-10-01 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 1 year
  Clinical pregnancy was confirmed by detection of one or more gestational sacs during transvaginal scan 4 weeks after embryo transfer.

SECONDARY OUTCOMES:
Follicle growth | 1 year
  Detection of estrogen level elevation and follicle diameter increases reflecting follicle growth.

CONTACTS AND LOCATIONS:
Overall Officials: Yingpu Sun, MD,PhD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhai J, Yao G, Dong F, Bu Z, Cheng Y, Sato Y, Hu L, Zhang Y, Wang J, Dai S, Li J, Sun J, Hsueh AJ, Kawamura K, Sun Y. In Vitro Activation of Follicles and Fresh Tissue Auto-transplantation in Primary Ovarian Insufficiency Patients. J Clin Endocrinol Metab. 2016 Nov;101(11):4405-4412. doi: 10.1210/jc.2016-1589. Epub 2016 Aug 29. PMID 27571179
- [Background] Donnez J, Martinez-Madrid B, Jadoul P, Van Langendonckt A, Demylle D, Dolmans MM. Ovarian tissue cryopreservation and transplantation: a review. Hum Reprod Update. 2006 Sep-Oct;12(5):519-35. doi: 10.1093/humupd/dml032. Epub 2006 Jul 18. PMID 16849817
- [Background] Li J, Kawamura K, Cheng Y, Liu S, Klein C, Liu S, Duan EK, Hsueh AJ. Activation of dormant ovarian follicles to generate mature eggs. Proc Natl Acad Sci U S A. 2010 Jun 1;107(22):10280-4. doi: 10.1073/pnas.1001198107. Epub 2010 May 17. PMID 20479243
- [Background] Kawamura K, Cheng Y, Suzuki N, Deguchi M, Sato Y, Takae S, Ho CH, Kawamura N, Tamura M, Hashimoto S, Sugishita Y, Morimoto Y, Hosoi Y, Yoshioka N, Ishizuka B, Hsueh AJ. Hippo signaling disruption and Akt stimulation of ovarian follicles for infertility treatment. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17474-9. doi: 10.1073/pnas.1312830110. Epub 2013 Sep 30. PMID 24082083